CLINICAL TRIAL: NCT06204133
Title: Model Study on Cervical Cancer Screening Strategies and Risk Prediction
Status: Completed | Type: Observational
Sponsor: Fujian Maternity and Child Health Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CSRM2304
Record Dates: First submitted 2023-12-15; First posted 2024-01-12 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Cervical Cancer Screening; Risk Assessment; Artificial Intelligence; Machine Learning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Artificial intelligence model building — Using non-image medical data of cervical lesions and clinical pathology results in different medical institutions, machine learning is adopted to establish multiple multi-modal cervical cancer intelligent screening prediction models. This method was used to analyze the prediction performance of the multi-modal cervical cancer intelligent screening prediction and risk triage model, and to evaluate and optimize the self-learning ability of the established multi-modal cervical cancer intelligent screening prediction model.

SUMMARY:
By collecting non-image medical data of women undergoing cervical screening in multiple centers in China, including age, HPV infection status, HPV infection type, TCT results, and colposcopy biopsy pathology results, a multi-source heterogeneous cervical lesion collaborative research big data platform was established. Based on artificial intelligence (AI) machine learning, cervical lesion screening features are refined, a multi-modal cervical cancer intelligent screening prediction and risk triage model is constructed, and its clinical application value is preliminarily explored.

DETAILED DESCRIPTION:
By collecting non-image medical data of women undergoing cervical screening in multiple centers in China, including age, HPV infection status, HPV infection type, TCT results, and colposcopy biopsy pathology results, a multi-source heterogeneous cervical lesion collaborative research big data platform was established. Based on artificial intelligence (AI) machine learning, cervical lesion screening features are refined, a multi-modal cervical cancer intelligent screening prediction and risk triage model is constructed, and its clinical application value is preliminarily explored. The effect of clinical application of the model was evaluated by internal data from Fujian Province and external data from several other regions in China.

ELIGIBILITY:
Inclusion Criteria:

* Age 25-64 years old;
* There was no history of precancerous lesions or cervical cancer;
* No previous cervical surgery or cervical removal;

Exclusion Criteria:

* HPV test results are not available;
* Pregnant or lactating women;
* There is a serious immune system disease, and the disease is active;

Ages: 25 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: For women aged 25-64 years who undergo cervical cancer screening, all women use HR-HPV testing as a primary screening strategy.
Sampling Method: Probability Sample
Enrollment: 1112846 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Cervical histopathology | within 8 weeks，
  Cervical histopathological diagnosis within 8 weeks
colposcopy | Percentage of patients diagnosed with cervical intraepithelial neoplasia of grade 3 (CIN3) or worse by cervical histopathological measurements within 8 weeks
  Colposcopists use colposcopic equipment to investigate the occurrence of cervical and vaginal lesions within 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pengming Sun, Study Chair — Fujian Maternal and Child Health Hospital
Locations (7):
- China (7):
  - Fujian Maternity and Child Health Hospital, Fuzhou, Fujian
  - Ningde maternal and child health hospital, Ningde, Fujian
  - Gansu Provincial Maternity and Child-care Hospital, Lanzhou, Ganshu
  - Shunde Women's and Children's Hospital of Guangdong Medical University, Foshan, Guangdong
  - Shenzhen Maternal and Child Health Hospital, Shenzhen, Guangdong
  - Guiyang maternal and child health care hospital, Guiyang, Guizhou
  - Hubei Maternal and Child Health Hospital, Wuhan, Hubei